CLINICAL TRIAL: NCT03464656
Title: Oxidative Stress In Semen And Male Infertility
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Fairhaven Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16351/16
Record Dates: First submitted 2018-02-26; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-01

CONDITIONS: Antioxidants; Infertility, Male; Semen Quality
Keywords: semen; male infertility; semen quality; sperm DNA fragmentation; oxidation reduction potential
MeSH Terms: conditions — Infertility, Male | interventions — Menogaril; Antioxidants; Semen Analysis; Seeds; Oxidative Stress

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, comparative study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients presenting with male infertility, who are found to have abnormal semen analysis shall be recruited to this study.
  Interventions:
  * Patients will be given Fairhaven Pro for Men as antioxidant in a dose of 3 tablets twice daily for 3 months.
  * Full assessment of fertility will be done.
  Interventions: Drug: Fairhaven Pro for men; Diagnostic Test: Semen analysis; Diagnostic Test: Sperm DNA fragmentation; Diagnostic Test: Static Oxidation reduction potential in semen

INTERVENTIONS:
Drug: Fairhaven Pro for men — Fairhaven Pro for men
  The antioxidant formula (Fairhaven Health) contains:
  * B12 (1000 mcg)
  * Zinc (30 mg)
  * Selenium (140 mcg)
  * Arginine (350 mg)
  * L-carnitine tartrate (2000 mg) , providing 1,340 mg of L-carnitine
  * CoQ10 (200 mg)
  * Vitamin C (120 mg) and Vitamin E (200 IU)
  Other Names: Antioxidant
Diagnostic Test: Semen analysis — Full semen analysis according to WHO semen laboratory manual 5th edition will be done pre and 3 months post-treatment.
  After complete liquefaction, each sample was evaluated for both macroscopic parameters such as color, pH, ejaculate volume, age of the sample and viscosity. An aliquot of the sample was examined for sperm concentration, total sperm count, total and progressive motility and sperm morphology using the WHO fifth edition guidelines (WHO, 2010). Semen analysis was done manually using a hemocytometer. Sperm motility was assessed and categorized as progressive or non-progressive. Morphology was assessed by a single experienced technician using the Diff-Quik staining protocol. Kruger's strict criteria were used for morphology assessment with 4% normal morphology as a cut-off (WHO, 2010).
  Other Names: Semen test
Diagnostic Test: Sperm DNA fragmentation — Sperm DNA fragmentation was evaluated using the Halosperm kit from Halotech DNA, S.L. (Madrid, Spain) as per manufacturer instructions. The method is based on the sperm chromatin dispersion test (Fernández et al., 2003). A minimum of 500 spermatozoa were scored and reported as percentage of sperm with spermatozoa with fragmented DNA. Normal value is measure at a cut-off value of more than 30%
  Other Names: SDF
Diagnostic Test: Static Oxidation reduction potential in semen — Oxidative stress was assessed by measuring the static oxidation-reduction potential (sORP) of neat liquefied semen samples using the MiOXSYSTM System (Aytu Bioscience, Inc., Englewood, USA). This is a galvanostatic measure of the electron transfer from reductants (antioxidants) to oxidants under a steady low voltage reducing current. Thus, providing an aggregate measure of all current oxidant activity and antioxidant activity in a sample. Higher sORP values (millivolts, mV) indicate a higher oxidant activity relative to the antioxidant activity and therefore greater state of oxidative stress.
  Other Names: sORP; Oxidative stress

SUMMARY:
The proposed research aims to study the effects of antioxidant therapy, commonly used in male infertility treatment, on semen analysis. Patients presenting with male infertility, who are found to have abnormal semen analysis shall be recruited to this study. They will be asked to provide a sample of semen for routine semen analysis and advanced semen tests including sperm DNA fragmentation and sORP before starting with antioxidant therapy and after 3-month treatment with antioxidants.

After completing the data analysis, we intend to publish the study in high impact perr reviewed journals and present it in international conferences.

DETAILED DESCRIPTION:
The proposed research aims to study the effects of antioxidant therapy, commonly used in male infertility treatment, on semen analysis. Several studies have been conducted to evaluate the effect of many antioxidant regimens on male infertility. A randomized double-blind, placebo-controlled trial investigated a combined antioxidant regimen, including vitamin C, using Menevit (lycopene 6mg, vitamin E 400IU, vitamin C 100mg, zinc 25mg, selenium 26 mcg, folate 0.5mg, garlic 1g) in couples undergoing intracytoplasmic sperm injection. The authors reported a significant improvement in viable pregnancy rate in the treatment group, where 38.5% of transferred embryos resulted in a viable fetus compared to 16% in the placebo group (Tremellen K, 2007). Suleiman et al. studied 300 mg of daily vitamin E in a placebo-controlled study revealing significant improvement in sperm motility and reduction of oxidative stress measures in the treatment group. Moreover, they reported a 21% spontaneous pregnancy rate in the treatment group compared to 0% in the placebo group (Suleiman SA, 1996).

Patients presenting with male infertility, who are found to have abnormal semen analysis shall be recruited to this study. They will be asked to provide a sample of semen for routine semen analysis and advanced semen tests including sperm DNA fragmentation and sORP before starting with antioxidant therapy and after 3-month treatment with antioxidants. No other procedures will be done for research purposes. All other investigations or treatments will be given according to the standard of care. Routinely patients presenting to the male infertility unit at HMC seeking evaluation and treatment for delayed conception will be assessed with a history and physical examination, investigated with semen and endocrine studies and be placed on an antioxidant regimen comprised of vitamins C and E, L-Carnitine and pentoxyfylline. Further management will be individualized and planned according to each patient's condition.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal sperm parameters defined as having at least two out of the following three criteria:
* Sperm Concentration > 1 and ≤ 15 million per ml
* Sperm total Motility ≤ 40%
* Sperm Morphology by Strict Criteria; normal forms ≤ 4.0%
* Absence of infection in semen (pus cells < 1 X 106/ml)
* No history of taking any therapy for their infertility including OTC treatment and vitamin supplementation
* No history of obstructive azoospermia
* No history of testicular cancer

Exclusion Criteria:

* Semen volume ≤ 1.5 mL
* Hydrocele, clinical varicocele (grade 2 and higher), orchitis, epididymitis, Cryptorchidism, irradiation or subjects that received chemotherapy treatment
* Clinically meaningful endocrinopathy defined as an endocrinopathy which requires endocrine medications (e.g. Diabetes, Thyroid disease, Pituitary diseases, Adrenal diseases, etc.) or measurement of the following hormonal values:

  1. Testosterone < 10.4 nmol/L
  2. LH <1 or > 9 IU/L and or FSH <1 or >19 IU/mL
  3. Elevated prolactin >407 mIU/L
  4. Elevated TSH > 4.5 U/mL
  5. Elevated Estrogen> 275 pmol/L
* Leukocytospermia: WBC count of > 1 X 106/ ml
* Known HIV infection
* Use of antioxidant agents or vitamins within 8 weeks prior to inclusion into the study
* Consumption of more than 1 unit of alcohol daily*
* Subjects following any special diet including, but not limited to liquid, high or low protein, raw food, vegetarian or vegan, etc.
* History of current use of illegal or "recreational" drugs
* History of malignancy not curatively treated at least 5 years before screening visit with exception of basal cell carcinoma in situ which may have been curatively treated within 1 year
* Participation in another clinical trial within 30 days or 7 half-lives of the prior test product, whichever is longer
* Any condition which, in the opinion of the investigator, might put the subject at risk by participation in this study

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of antioxidant therapy on sperm motility in infertile men, | 1 year
  Measured by mean change in sperm motility pre- and post-treatment with antioxidants.
Evaluate the effect of antioxidant therapy on sperm morphology in infertile men | 1 year
  Measured by the mean change in sperm morphology pre- and post-treatment with antioxidants
Evaluate the effect of antioxidant therapy on sperm count in infertile men | 1 year
  Measured by mean change in sperm count pre- and post-treatment with antioxidants.

SECONDARY OUTCOMES:
Evaluate the effect of antioxidant therapy on sperm DNA fragmentation in infertile men | 1 year
  Difference in mean change in sperm DNA fragmentation pre and post-treatment
Evaluate the effect of antioxidant therapy on oxidative stress in infertile men | 1 year
  Measure difference in mean change in seminal oxidation reduction potential in infertile men pre- and post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar